CLINICAL TRIAL: NCT04399122
Title: Post-operative Pain Control After Photorefractive Keratectomy Comparing Acetaminophen/Codeine vs Acetaminophen/Oxycodone
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: 59th Medical Wing (U.S. Federal Agency)
Responsible Party: Principal Investigator, Charisma Evangelista, Chief of Refractive Surgery, 59th Medical Wing
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: FWH20160007H
Record Dates: First submitted 2020-05-19; First posted 2020-05-22 (Actual); Results first posted 2021-10-05 (Actual); Last update posted 2021-10-05 (Actual); Status verified 2021-09

CONDITIONS: Post-operative Pain Control
Keywords: Photorefractive Keratectomy; Post-operative Eye Pain; Refractive Surgery
MeSH Terms: interventions — Acetaminophen

STUDY DESIGN:
Intervention Model Description: Patients will be randomized to Group 1 or Group 2
Who Masked: Participant, Investigator
Masking Description: Randomization was accomplished by the pharmacy and the medication bottles were not labeled.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Acetaminophen with codeine (Active Comparator): codeine 30mg/acetaminophen 325mg Take one to two tablets every 4 to 6 hours as needed for pain for up to 4 days following surgery.
  Interventions: Drug: acetaminophen/codeine vs acetaminophen/oxycodone
- Acetaminophen with oxycodone (Active Comparator): oxycodone 5mg/acetaminophen 325mg Take one tablet every 4 to 6 hours as needed for pain for up to 4 days following surgery.
  Interventions: Drug: acetaminophen/codeine vs acetaminophen/oxycodone

INTERVENTIONS:
Drug: acetaminophen/codeine vs acetaminophen/oxycodone — pain medications
  Other Names: Tylenol 3 VS Percocet

SUMMARY:
Photorefractive keratectomy (PRK) is a refractive error correction procedure that helps eliminate or reduce the dependence on corrective lenses. An important aspect of PRK is post-operative pain management. Post-operative pain can be significant in the first three to five days and is typically controlled utilizing various modalities including narcotic pain medication. Simple observation suggests a difference in the post-operative pain levels of patients utilizing the more potent oxycodone- versus the less potent codeine-containing acetaminophen preparations. There have been no studies performed to explore any differences in perceived pain comparing these two medications when used following PRK. This study is designed to answer this question by means of a pain survey conducted in the first five days post-op. This may help better manage similar patients in the future.

DETAILED DESCRIPTION:
This will be a prospective pain assessment study utilizing a simple three question survey given to patients undergoing bilateral PRK. Following recruitment and enrollment (see section 4.1 and 4.2 for recruitment and consent process), patients will be randomized to be prescribed either 1) Group 1: codeine 30mg/acetaminophen 300mg (standard of care dosage) or 2) Group 2: oxycodone 5mg/acetaminophen 325mg (standard of care dosage) post-operatively. All post-operative patients will receive standard bandage contact lenses and as needed tetracaine as per standard of care. Patients will be removed from the study if they take other non-study pain medications. They will be asked to record their pain levels four times daily as well as the number of as needed narcotic pain medication taken and the number of tetracaine drops used (to isolate a potential confounding pain control modality). Randomization will be performed with the aid of www.randomizer.org which will generate a randomized assignment to either group 1 or group 2.

All PRK procedures will be performed per standard of care. The procedure will be performed by one of the 4 approved surgeons. All surgeons will use the same technique using either the VISX or the Allegretto laser machines. This technique will include use of a brush for mechanical removal of corneal epithelial cells. The surgeons will take note at this time of the relative adherence of the epithelium to the underlying tissue and grade the adherence on a scale of 0-4 (0=least adherent and 4=most adherent). In the data analysis, differences between surgeons and between operating platform (VISX vs Allegretto) will be compared to account for any possible bias in operating parameters.

The survey will be worded as follows:

1. "Rate your eye pain or level of discomfort at 0800, 1200, 1600 and 2000. Please write the number closest to your response in the table below under the appropriate day and time.
2. "How many tablets of study-related pain medication did you take today in the AM/PM?"
3. "How many times did you use topical tetracaine today in the AM/PM?"
4. "Did you take any other non-study related pain medications?"

Patients will be followed-up post-operatively as per standard of care. This includes follow-up visits at 1 day, 1 week, 1 month, 3 months, 6 months and 12 months. Starting on post-operative day 1, the patients will be asked to record their pain levels using the pain survey at four hour intervals (0800, 1200, 1600, 2000). At the 1 week post-operative visit, the pain surveys will be collected from the patients. Visual acuity data will be extracted from all but the 12 month follow-up appointment and used as a secondary outcome to correlate any possible differences in pain scores to functional outcomes in terms of visual acuity.

ELIGIBILITY:
Inclusion Criteria:

* M/F >21 years of age (PRK is not done on anyone under the age of 21 at this surgery center)
* Have met all criteria for bilateral PRK

Exclusion Criteria

* Patients who do not meet the criteria for refractive surgery
* Patients receiving LASIK
* Patients known to have an allergy to either of the study pain medications
* Patients receiving refractive surgery on only one eye
* Pregnant women, children, military basic trainees, prisoners and detainees
* Subject has used narcotics in the last 6 months

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2017-03-21 (Actual); Primary Completion 2019-10-28 (Actual); Study Completion 2019-10-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charisma B Evangelista, MD, Principal Investigator — 59th Medical Wing
Locations (1):
- Joint Warfighter Refractive Surgery Center at WHASC, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: In this single-center, double-masked randomized clinical trial, patients were recruited at the Joint Warfighter Refractive Surgery Center (JWRSC) at Wilford Hall Ambulatory Surgical Center, Lackland Air Force Base, Texas, between March 2016 and April 2019.
Period: Overall Study
Arm/Group | Acetaminophen With Codeine | Acetaminophen With Oxycodone
Started | 100 | 100
Completed | 97 | 100
Not Completed | 3 | 0
Not completed — Lost to Follow-up | 2 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Population: Three participants withdrew from the acetaminophen with codeine arm: One participant withdrew from the study because they did not wish to proceed with refractive surgery. Two participants withdrew due to their inability to return for all required follow-up visits.
Groups:
- Total: Total of all reporting groups
Arm/Group | Acetaminophen With Codeine | Acetaminophen With Oxycodone | Total
Number analyzed (Participants) | 97 | 100 | 197
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 97 | 100 | 197
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.5 (7.5) | 31.5 (6.5) | 32.5 (6.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 81 | 73 | 154
  Male | 16 | 27 | 43
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 97 | 100 | 197

OUTCOME MEASURES:

1. Primary Outcome: Post-operative Average Pain Score
Description: The PRK Post-Operative Pain Survey consisted of a scale of 0 - 10 with a score of 0 equal to no pain, a score of 1 - 3 equal to mild pain, a score of 4 - 6 equal to moderate pain and a score of 7 - 10 equal to severe pain
Time Frame: 2 days post surgery
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Acetaminophen With Codeine | Acetaminophen With Oxycodone
Number analyzed (Participants) | 97 | 100
units on a scale | 2.82 (2.03) | 3.58 (2.29)

2. Secondary Outcome: Post-operative Uncorrected Visual Acuity Right and Left Eye
Description: Right and left eye uncorrected visual acuity at post-operative month 6.
Time Frame: Post-operative month 6.
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | Acetaminophen With Codeine | Acetaminophen With Oxycodone
Number analyzed (Participants) | 97 | 100
logMAR
  Right Eye logMAR | -0.07 (0.01) | -0.05 (0.01)
  Left Eye logMAR | -0.06 (0.01) | -0.06 (0.01)

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Acetaminophen With Codeine | Acetaminophen With Oxycodone
All-Cause Mortality (participants affected / at risk) | 0/97 | 0/100
Serious Adverse Events (participants affected / at risk) | 0/97 | 0/100
Other Adverse Events (participants affected / at risk) | 0/97 | 0/100

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2017-09-06): https://cdn.clinicaltrials.gov/large-docs/22/NCT04399122/Prot_001.pdf